CLINICAL TRIAL: NCT04877210
Title: Effects of Topical Insulin on Levels of Tear Inflammatory Mediators Compared to Standard Artificial Tears and Normal Saline in Diabetics With Dry Eye Disease
Brief Title: Effects of Topical Insulin on Levels of Tear Inflammatory Mediators
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Mae-Lynn Catherine Bastion, Professor Dr, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PPUKM
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical Insulin (Experimental): Insulin (Actrapid) diluted in normal saline
  Interventions: Drug: Topical Insulin
- Normal Saline (Placebo Comparator): Normal saline eyedrops
  Interventions: Drug: Topical Insulin
- Standard Artifical Tear (Active Comparator): Gutt systane ultra
  Interventions: Drug: Topical Insulin

INTERVENTIONS:
Drug: Topical Insulin — Insulin (Actrapid) diluted in Normal Saline is given to participant 1 drop to both eyes 4 times per days for 4 weeks
  Other Names: Gutt insulin

SUMMARY:
60 samples are take to determine the effects of topical insulin on tear inflammatory mediators interleukin 1a, interleukin 6 and matrix metalloprotenase 9 in diabetics with dry eye disease.

DETAILED DESCRIPTION:
Tear samples are taken to compare the levels of inflammatory markers (IL 1a, IL6 and MMP 9) pre-and post treatment with topical insulin in normal saline compared to standard therapy and normal saline in diabetics with dry eyes and also to correlate the IL 1a, IL6 and MMP 9 levels with clinical outcomes in diabetics with dry eyes treated with topical insulin in normal saline, standard therapy and normal saline

ELIGIBILITY:
Inclusion Criteria:

* all diabetics aged 18 - 50 years of age with at least mild OSDI scores

Exclusion Criteria:

* Diabetics on contact lenses
* Diabetic with history of ocular surgery in the preceding 3 months
* Post menopausal women
* Known mild dry eye with prior usage of topical therapy who are unable to discontinue
* Known case of allergic eye disease
* Sjogren's syndrome patients
* Unwilling or unable to attend 6 follow up and sampling sessions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-01-26 (Estimated)

PRIMARY OUTCOMES:
Biochemical marker 1 | 4 weeks
  Interleuikn 1-alpha
Biochemical marker 2 | 4 weeks
  Interleukin 6
Biochemical marker 3 | 4 weeks
  Matrix metallo-proteinase 9

CONTACTS AND LOCATIONS:
Overall Officials: Mae-Lynn C. Bastion, Principal Investigator — PPUKM
Locations (1):
- PPUKM, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes